CLINICAL TRIAL: NCT05108207
Title: Software-guided Cognitive Stimulation Prevents the Development of Delirium in Hospitalized Older Adults: Randomized Controlled Trial
Brief Title: A Software to Prevent Delirium (PREVEDEL) in Hospitalized Older Adults
Acronym: PREVEDEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Tobar, Eduardo Tobar, Associated professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ID16AM2080
Record Dates: First submitted 2021-08-05; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Delirium; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations
Keywords: delirium; prevention; cognitive stimulation
MeSH Terms: conditions — Delirium; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations

STUDY DESIGN:
Intervention Model Description: Multi-center, parallel-group, randomized controlled trial (RCT). CONSORT methodological recommendations are used for reporting non-pharmacological trials, in addition to TIDieR and SPIRIT recommendations.
Who Masked: Outcomes Assessor
Masking Description: The enrollers, evaluators and healthcare personnel (nurses, physical therapists, physicians, occupational therapists) do not know the assigned group. Both groups receive a tablet of the same dimensions and with the same basic applications. However, blinding the patient is not possible, since when exploring the tablet, he or she will recognize whether or not it has the PREVEDEL program included. To reduce this bias, the staff that delivers the tablet encourages both groups to use its different basic applications (access the Internet) and that any doubts may have participants about its use should be made to the tablet coordinator, so that the evaluators or healthcare personnel remain masked.
  The time between assignment and delivery of the tablet is between 4 to 12 hours in all participating centers. This variable will be measured for later analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): will receive the standard delirium prevention measures outlined above, plus the use of a mobile device without delirium prevention software for 5 days (Control Group: nPPD package, without PREVEDEL).
  Interventions: Other: Placebo; Other: Implement a program of non-pharmacological interventions to prevent delirium
- Experimental Group (Experimental): will receive the standard delirium prevention measures, plus the use of a mobile device with PREVEDEL software for 5 days (Experimental Group: nPPD package, with PREVEDEL).
  Interventions: Other: Prevention software; Other: Implement a program of non-pharmacological interventions to prevent delirium

INTERVENTIONS:
Other: Prevention software — The software is installed on an Alcatel OneTouch Pixi-3 10 tablet and is delivered every day to each patient between 9:00 am and 8:00 pm, with nighttime pickup (8:00 pm to 09:00 am), so the patient can rest and to charge the device. The first day, a previously trained health professional delivers the tablet and trains the older adults in its use, taking 10 to 15 minutes. The day after the tablet is delivered, the same person goes to the patient's room to check if he or she has any doubts or problems with its use. Both groups are advised to use the tablet 3 times a day, at least 10 minutes each time.
  Arms: Experimental Group
Other: Placebo — All patients will have a tablet without the software PREVEDEL between 09:00-19:00 hrs.
  Arms: Control Group
Other: Implement a program of non-pharmacological interventions to prevent delirium — Three months before the start of the clinical trial, an intervention is carried out in the Internal Medicine, Geriatrics and Intermediate Care Unit services of the 4 participating centers in order to establish a homogeneous plan of nPPD and assess adherence. The implementation methodology in the first stage will be according to the Consolidated Framework for Advancing Implementation Science (CFIR) model, used in a local pilot study.

SUMMARY:
Background

Delirium, is a clinical condition characterized by acute and fluctuating deterioration of the cognitive state, generally secondary to an acute pathology. It is a common condition in hospitalized older adults and it develops in 20-30% of patients hospitalized in a general ward and up to 80% of those hospitalized in critical care units. Delirium is associated with negative outcomes in older adults, such as longer hospitalizations, higher mortality, and short and medium-term institutionalization. Randomized clinical trials have shown that delirium is preventable through non-pharmacological prevention measures, decreasing its incidence by 30 to 50%. These interventions include promoting physical activity, facilitating the use of glasses and hearing aids, cognitive stimulation, and providing frequent reorientation of time and space, among others.

These measures are currently seldom applied in hospitals in Chile and around the world for various reasons some of which include the heavy workload of clinical staff, the lack of trained personnel, and, in general, the absence of systematic implementation processes.

The main objective is to evaluate whether cognitive stimulation guided by PREVEDEL software prevents delirium status(full/subsyncromal delirium) in hospitalized older adults.

Method/Design: randomized controlled trial, parallel groups, multicenter.

Participants: patients 65 years or older who have been hospitalized for less than 48 hours in the general ward or in the intermediate care unit of 4 hospitals in Santiago, Chile.

Intervention: participants in the intervention group will use a tablet with cognitive stimulation software for delirium prevention for 5 continuous days versus the control group who will use the tablet without the software.

Evaluations: The incidence of delirium and subsyndromal delirium, duration, density of delirium, cognitive and functional status at discharge, adherence to prevention measures, as well as demographic variables of interest will be evaluated.

DETAILED DESCRIPTION:
Background. Delirium is a clinical condition characterized by acute cognitive impairment, of fluctuating course, generally secondary to an acute pathology, which appears after the interaction between predisposing factors and well described precipitants. It is a very common condition in older adults, observed in 20% to 30% of patients hospitalized in a general ward, and up to 80% of those hospitalized in critical care units. Delirium is associated with negative clinical outcomes which include longer hospitalizations, increased direct and indirect costs, functional impairment, greater risk of mortality, increased risk of institutionalization, and deterioration in long-term cognitive status, among others.

Subsyndromal delirium (SSD) is a milder state characterised by the presence of certain delirium symptoms but without meeting full diagnostic criteria thresholds, is also associated with poor posthospitalization outcomes similar to those associated with delirium. The reported frequency of subsyndromal delirium varies (7-50%) according to the definition applied and the clinical population studied. Its incidence in the general medicine ward is 17%.

The frequency of delirium status (full/subsyndromal delirium) in the general room is approximately 25%.

It is known that delirium in hospitalized older adults is preventable. In multiple randomized clinical trials, non-pharmacological interventions to prevent delirium (nPPD), shown to reduce its incidence by 30-50%7.

Despite the high evidence supporting them, non-pharmacological interventions to prevent delirium are poorly implemented in hospitals in Chile and around the world for several reasons, such as the heavy workload of clinical staff, lack of trained personnel, and, in general, the absence of systematic implementation processes.

Prior to this clinical trial, local pilot studies have shown some progress in this area. On the one hand, it has been reported that the incorporation of software technology through a "PREVEDEL" tablet is feasible and can be implemented on a hospital level, with possible effects on decreasing delirium. On the other hand, the implementation of nPPD following a theoretical model improves the adherence of health personnel.

Therefore, a multicenter randomized clinical trial is proposed, which seeks to evaluate whether cognitive stimulation guided by the PREVEDEL software prevents delirium in hospitalized older adults and whether it is a technology that can be used in others hospital centers.

Centers and place where data is collected. Chile. These are: Hospital Clínico de la Universidad de Chile (HCUCH), Hospital San Juan de Dios (HSJD), Clínica Las Condes (CLC) and Hospital Santiago Oriente Dr. Luis Tisné (HLT). Two are public institutions and two are private institutions.

Intervention.

Interventions to implement a program of non-pharmacological interventions to prevent delirium (nPPD) in the centers that will participate in the RCT.

Three months before the start of the clinical trial, an intervention is carried out in the Internal Medicine, Geriatrics and Intermediate Care Unit services of the 4 participating centers in order to establish a homogeneous plan of nPPD and assess adherence. The implementation methodology in the first stage will be according to the Consolidated Framework for Advancing Implementation Science (CFIR) model, used in a local pilot study

Interventions to perform an RCT where the effect of the use of PREVEDEL versus a placebo (Tablet without PREVEDEL) in the prevention of delirium in older adults is compared.

Standard non-pharmacological prevention measures

According to the recommendations in the literature and those made by local studies, the following standard non-pharmacological delirium prevention measures were defined:

Study groups Control Group: will receive the standard delirium prevention measures outlined above, plus the use of a mobile device without delirium prevention software for 5 days (Control Group: nPPD package, without PREVEDEL).

Experimental Group: will receive the standard delirium prevention measures, plus the use of a mobile device with PREVEDEL software for 5 days (Experimental Group: nPPD package, with PREVEDEL).

To evaluate patient adherence and how the tablet is used, both groups will have an application installed in their devices that will allow them to keep track of the time of use and applications used.

Software content

1. Desktop module.
2. The exercise module.
3. Games module.
4. The documentary module.
5. Alert module.
6. Configuration module, allows software customization.
7. Registration system.

OBJECTIVES AND HYPOTHESIS

General To assess whether cognitive stimulation guided by PREVEDEL software prevents delirium status in hospitalized older adults.

Specifics

* Implement a program of nPPD at the centers that will participate in the randomized clinical trial (RCT).
* Conduct a randomized clinical trial (RCT) comparing the effect of the use of PREVEDEL versus placebo (Tablet without PREVEDEL) in the prevention of delirium in older adults.

Hypothesis Cognitive stimulation guided by PREVEDEL software decreases the incidence of delirium status in hospitalized older adults.

Study sample.

For the calculation of the sample size, local and literature data were considered. A delirium status prevalence of 20% is estimated in the Control group and a decrease of this to 8% in the Intervention group. In this way, with a power of 80%, and an alpha of 0.05 bilaterally, 147 patients will be enrolled in each group. If add to this a 10% loss of follow-up, the overall sample size is 320 patients.

Randomization. Randomization was performed with computer-generated random permuted blocks using a centralized, secure Web-based randomization service.

Masking The enrollers, evaluators and healthcare personnel (nurses, physical therapists, physicians, occupational therapists) do not know the assigned group. Both groups receive a tablet of the same dimensions and with the same basic applications. However, blinding the patient is not possible, since when exploring the tablet, he or she will recognize whether or not it has the PREVEDEL program included. To reduce this bias, the staff that delivers the tablet encourages both groups to use its different basic applications (access the Internet) and that any doubts may have participants about its use should be made to the tablet coordinator, so that the evaluators or healthcare personnel remain masked.

The time between assignment and delivery of the tablet is between 4 to 12 hours in all participating centers. This variable will be measured for later analysis.

Statistical Methods For the descriptive analysis of the variables will use the mean (standard deviation), median (25-75 percentiles), or proportions as appropriate to the type and distribution of the data.

Analytical Statistics: For the primary outcome, a comparison of proportions between patients who develop delirium and subsyndromal delirium in both groups will be made, using Fisher's exact test, and as a measure of efficacy, an OR (95% CI) will be estimated. If there is any baseline variable that is not matched by the randomization, efficacy analyses will be carried out by means of logistic regression with the main variable being the treatment, and the adjustment variables those that the randomization would not have been able to match. Additionally, to compare the effect of the intervention over time, a time-to-event analysis will be performed using the Kaplan-Maier procedure and then the Cox regression model to adjust for baseline variables and the presence of the intervention. For the secondary outcomes, the Fisher's exact test or t-Test will be used, as appropriate, for the type and distribution of the data. Linear regression or multivariate logistics will also be performed, as appropriate, to evaluate the impact of the intervention, adjusting for the input covariates. A bilateral p 0.05 significance level will be used for all analyses.

Ethics Committee The research protocol was reviewed and approved by the ethics committee of the Clinical Hospital of the University of Chile and its approval was validated by the ethics committees of the respective participating centers (Registry No. 049, July 31, 2019).

Trial Steering Committee

Committee was formed with 3 international experts in the "Trial Steering Committee" (TSC) area. This committee will watch over the following aspects:

* Supervise and guarantee scientific quality.
* Advise on study protocol, recruitment progress, adherence, follow-up and data quality.
* Review the recommendations of the data analysis and monitoring committee.
* Review the publications in the primary trials.

For the fulfillment of the objectives, the TSC will meet before, in the middle and at the end of the recruitment.

Informed Consent The informed consent will be given by the patient himself and obtained by one of the main investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years or older.
* Hospitalized less than an 48 hours ago in a general ward or in the intermediate care unit. Participating health center: 1) Hospital Clínico de la Universidad de Chile, 2) Hospital San Juan de Dios, 3) Clínica Las Condes, 4) Hospital Santiago Oriente Dr Luis Tisné.

Exclusion Criteria:

* Presence of full or syndromal delirium (CAM+ or presence of one core elements).
* History of dementia (AD8 greater than 2 points).
* Non-Spanish speaking patients.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Delirium Status (delirium and subsyndromal delirium) | 5 days
  To evaluate the incidence of delirium and incidence of subsyndromal with Confusion Assessment Method (CAM).

SECONDARY OUTCOMES:
Duration of delirium | 5 days of protocol and 2 days of follow-up.
  To evaluate duration in days.
Density of delirium | 5 days.
  Understood as the ratio between the duration of the event and the exposure time (time spent in the protocol).
Level of independence in basic activities of daily living | At day 0 and 5.
  To evaluate level of independence in activities of daily living at discharge with Functional Independence Measure.Scoring ranges from 13 to 126 points, with higher scores indicative of better performance.
Cognitive level | At day 0 and 5.
  Evaluate cognitive performance at hospital discharge with Montreal cognitive Assessment. Scoring ranges from 0 to 30 points, with higher scores indicative of better performance.
Adherence to prevention measures | At day 0 and 30 (before and after training in prevention measure).
  Assessment of adherence to 4 non-pharmacological prevention domains (12 indicators): Management of environment (visible clock, visible calendar, decrease physical restrictions, early mobilization), (indication of relative rest, encourage patient to sit and stand), correction of sensory deficits (availability of glasses, hearing aids, and dentures when necessary), management of medications (decrease the use of benzodiazepines, anticholinergics, and metoclopramide when possible).
Time of use of electronic device | 5 days
  The usage time on the mobile device (with internal device registration) will be recorded.
Hospital stay | Through study completion an average of 30 days
  Length of hospital stay in days.From the day of admission to the hospital until discharge.
90-day mortality | At 90 day.
  90-day mortality check by civil registry.
Difficulty falling and staying asleep due to device use. | Every day for 5 days.
  Every day when removing the device, the person will be asked ¿Have you had difficulty falling and staying asleep due to device use?
Headache due to the device use. | Every day for 5 days.
  Every day when removing the device, the person will be asked Have you had a headache due to the device use? If the answer is yes, the intensity of the pain will be scored, where 0 is no pain and 10 is the greatest pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Result] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Result] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Result] Veiga D, Luis C, Parente D, Fernandes V, Botelho M, Santos P, Abelha F. Postoperative delirium in intensive care patients: risk factors and outcome. Rev Bras Anestesiol. 2012 Jul;62(4):469-83. doi: 10.1016/S0034-7094(12)70146-0. PMID 22793963
- [Result] Leslie DL, Zhang Y, Holford TR, Bogardus ST, Leo-Summers LS, Inouye SK. Premature death associated with delirium at 1-year follow-up. Arch Intern Med. 2005 Jul 25;165(14):1657-62. doi: 10.1001/archinte.165.14.1657. PMID 16043686
- [Result] Sepulveda E, Leonard M, Franco JG, Adamis D, McCarthy G, Dunne C, Trzepacz PT, Gaviria AM, de Pablo J, Vilella E, Meagher DJ. Subsyndromal delirium compared with delirium, dementia, and subjects without delirium or dementia in elderly general hospital admissions and nursing home residents. Alzheimers Dement (Amst). 2016 Dec 1;7:1-10. doi: 10.1016/j.dadm.2016.11.002. eCollection 2017. PMID 28116342
- [Result] Meagher D, O'Regan N, Ryan D, Connolly W, Boland E, O'Caoimhe R, Clare J, Mcfarland J, Tighe S, Leonard M, Adamis D, Trzepacz PT, Timmons S. Frequency of delirium and subsyndromal delirium in an adult acute hospital population. Br J Psychiatry. 2014 Dec;205(6):478-85. doi: 10.1192/bjp.bp.113.139865. Epub 2014 Oct 30. PMID 25359923
- [Result] Abraha I, Trotta F, Rimland JM, Cruz-Jentoft A, Lozano-Montoya I, Soiza RL, Pierini V, Dessi Fulgheri P, Lattanzio F, O'Mahony D, Cherubini A. Efficacy of Non-Pharmacological Interventions to Prevent and Treat Delirium in Older Patients: A Systematic Overview. The SENATOR project ONTOP Series. PLoS One. 2015 Jun 10;10(6):e0123090. doi: 10.1371/journal.pone.0123090. eCollection 2015. PMID 26062023
- [Result] Inouye SK, Bogardus ST Jr, Charpentier PA, Leo-Summers L, Acampora D, Holford TR, Cooney LM Jr. A multicomponent intervention to prevent delirium in hospitalized older patients. N Engl J Med. 1999 Mar 4;340(9):669-76. doi: 10.1056/NEJM199903043400901. PMID 10053175
- [Result] Alvarez EA, Garrido MA, Tobar EA, Prieto SA, Vergara SO, Briceno CD, Gonzalez FJ. Occupational therapy for delirium management in elderly patients without mechanical ventilation in an intensive care unit: A pilot randomized clinical trial. J Crit Care. 2017 Feb;37:85-90. doi: 10.1016/j.jcrc.2016.09.002. Epub 2016 Sep 10. PMID 27660922
- [Result] Nydahl P, Dewes M, Dubb R, Hermes C, Kaltwasser A, Krotsetis S, von Haken R. Survey among critical care nurses and physicians about delirium management. Nurs Crit Care. 2018 Jan;23(1):23-29. doi: 10.1111/nicc.12299. Epub 2017 May 18. PMID 28523698
- [Result] Xing J, Sun Y, Jie Y, Yuan Z, Liu W. Perceptions, attitudes, and current practices regards delirium in China: A survey of 917 critical care nurses and physicians in China. Medicine (Baltimore). 2017 Sep;96(39):e8028. doi: 10.1097/MD.0000000000008028. PMID 28953621
- [Result] Alvarez EA, Garrido M, Ponce DP, Pizarro G, Cordova AA, Vera F, Ruiz R, Fernandez R, Velasquez JD, Tobar E, Salech F. A software to prevent delirium in hospitalised older adults: development and feasibility assessment. Age Ageing. 2020 Feb 27;49(2):239-245. doi: 10.1093/ageing/afz166. PMID 31957783
- [Result] Garrido MA, Alvarez EA, Ponce DP, Salech F, Tobar DI, Tobar EA. Consolidated framework for advancing implementation science for the implementation process and adherence assessment of a non-pharmacological delirium prevention program. Int J Geriatr Psychiatry. 2021 Feb;36(2):302-313. doi: 10.1002/gps.5425. Epub 2020 Sep 16. PMID 32892410
- [Result] Wei LA, Fearing MA, Sternberg EJ, Inouye SK. The Confusion Assessment Method: a systematic review of current usage. J Am Geriatr Soc. 2008 May;56(5):823-30. doi: 10.1111/j.1532-5415.2008.01674.x. Epub 2008 Apr 1. PMID 18384586
- [Result] Young Y, Fan MY, Hebel JR, Boult C. Concurrent validity of administering the functional independence measure (FIM) instrument by interview. Am J Phys Med Rehabil. 2009 Sep;88(9):766-70. doi: 10.1097/PHM.0b013e3181a9f1d6. PMID 19487922
- [Derived] Garrido M, Alvarez E, Salech F, Rojas V, Jara N, Farias JI, de la Vega DP, Tobar E. Software-guided (PREVEDEL) cognitive stimulation to prevent delirium in hospitalised older adults: study protocol. BMC Geriatr. 2023 Aug 5;23(1):472. doi: 10.1186/s12877-023-04189-2. PMID 37543590